CLINICAL TRIAL: NCT04119323
Title: Image Location and Performance of Left Bundle Branch Pacing
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: IMAGE-LBBP study
Record Dates: First submitted 2019-09-30; First posted 2019-10-08 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Cardiac Pacing; Pacing Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multi-site, non-randomized, data collection study. The purpose of this study is to investigate the correlation between pacing sites and ECG morphology or pacing parameters during left bundle branch pacing (LBBP) and perform the use condition analysis to assess the long-term performance of pacing lead during LBBP.

DETAILED DESCRIPTION:
His bundle pacing (HBP) is a physiological pacing, but also has some limitations, including high and unstable pacing threshold in 5-10% patients, low R-wave amplitude causing inappropriate pacing management, damage to the His bundle during implantation. On the other hand, left bundle branch pacing (LBBP), achieved via trans-ventricular septal approach with the pacing lead tip at the left side of the ventricular septum, has recently initiated and been widely practiced in China because of easy implantation, relatively narrow paced QRS duration, low and stable pacing threshold, high R wave amplitude, and the LBBB correction by a low pacing output.

As LBBP is in the early phase of clinical practice in China, in order to better conduct LBBP implantation and understand mechanisms of LBBP therapy, physicians often do imaging assessment of the pacing lead in patients implanted with LBBP based on clinical necessity.

Additionally, there is no report of mid/long-term correlation between lead location and ventricular electrical activity, nor mid/long-term pacing lead performance assessment during LBBP.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 80 years old;
* Patients providing signed Informed Consent;
* Patients indicated for permanent pacing and implanted with LBBP for at least 3 months, with documentation of implantation records;
* Patients who plan to receive cardiac CT examination.

Exclusion Criteria:

* Patients who have a history of allergy to contrast agent or refuse to use contrast agent in CT examination;
* Patients who are pregnant or have a plan for pregnancy during the study;
* Patients who are not willing to provide Informed Consent;
* Patients who have medical conditions that would limit study participation;
* Patients who were already enrolled in other clinical trial which would impact his/her participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for LBBP and implanted with pacing lead for LBBP.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
QRS duration | at least 3 months after implant
  The primary endpoint is QRS duration and morphology during LBBP

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Zhou, M.D., Study Director — Medtronic
Locations (3):
- China (3):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - West China Hospital, Chengdu, Sichuan

REFERENCES:
- [Derived] Cai M, Qiu Y, Xu Y, Lu H, Chen Z, Hou X, Jiang L, Zhou X, Dai Y, Liu X, Zou J, Chen K. Distance From Pacing Lead Tip to Left Ventricular Cavity Predicts Long-term Loss of Left Bundle Branch Capture: Insights From the IMAGE-LBBP Cohort. Can J Cardiol. 2025 Nov 1:S0828-282X(25)01291-7. doi: 10.1016/j.cjca.2025.10.032. Online ahead of print. PMID 41177376
- [Derived] Zou J, Chen K, Liu X, Xu Y, Jiang L, Dai Y, Lin J, Hou X, Qiu Y, Himes A, Lucas R, Demmer W, Mara N, Zhou X, Lu H. Clinical use conditions of lead deployment and simulated lead fracture rate in left bundle branch area pacing. J Cardiovasc Electrophysiol. 2023 Mar;34(3):718-725. doi: 10.1111/jce.15843. Epub 2023 Feb 14. PMID 36738153